CLINICAL TRIAL: NCT00080886
Title: A Phase II Trial Of BEAM/Rituximab/Autologous Hematopoietic Stem Cell Transplantation (AHSCT) For Patients With CD20 Positive Non-Hodgkin's Lymphoma
Brief Title: Rituximab, Carmustine; Cytarabine, Etoposide, & Melphalan; Stem Cell Transplantation for Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0063-02-FB; CDR0000357306 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Lymphoma
Keywords: recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Carmustine; Cytarabine; Etoposide; etoposide phosphate; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Other): Participants receive rituximab IV over approximately 3-4 hours once weekly for 2 weeks followed 1 week later by hematopoietic stem cell or bone marrow harvest.
  Participants then receive a third dose of rituximab IV over approximately 3-4 hours on day -7 or -6. Patients also receive high-dose chemotherapy comprising carmustine IV on day -6, cytarabine IV and etoposide IV twice daily on days -5 to -2, and melphalan IV on day -1. Participants undergo autologous hematopoietic stem cell transplantation on day 0. Participants who have less than a complete remission at day 100 post-transplantation receive 4 additional doses of rituximab IV over approximately 3-4 hours once weekly for 4 weeks. Participants are followed at day 100, at 1 year, and then annually thereafter.
  Interventions: Biological: rituximab; Drug: carmustine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: rituximab
  Other Names: Rituxan
Drug: carmustine
  Other Names: Gliadel Wafer, Bicnu
Drug: cytarabine
  Other Names: cytosine arabinoside
Drug: etoposide
  Other Names: Etopophos, Toposar
Drug: melphalan
  Other Names: Evomela
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as carmustine, cytarabine, etoposide, and melphalan, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining rituximab and combination chemotherapy with autologous stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining rituximab with combination chemotherapy followed by autologous hematopoietic stem cell transplantation in treating patients who have B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the levels of soluble CD20 antigen (sCD20) in the blood before and after treatment with rituximab and carmustine, cytarabine, etoposide, and melphalan followed by autologous hematopoietic stem cell transplantation in patients with CD20-positive B-cell non-Hodgkin's lymphoma.
* Correlate the effect of changes in levels of sCD20 with clinical outcomes in patients treated with this regimen.
* Determine the response rate in patients treated with this regimen.
* Determine the event-free survival of patients treated with this regimen.
* Determine the toxicity profile of this regimen in these patients.

OUTLINE: Patients receive rituximab IV over approximately 3-4 hours once weekly for 2 weeks followed 1 week later by hematopoietic stem cell or bone marrow harvest.

Patients then receive a third dose of rituximab IV over approximately 3-4 hours on day -7 or -6. Patients also receive high-dose chemotherapy comprising carmustine IV on day -6, cytarabine IV and etoposide IV twice daily on days -5 to -2, and melphalan IV on day -1. Patients undergo autologous hematopoietic stem cell transplantation on day 0.

Patients who have less than a complete remission at day 100 post-transplantation receive 4 additional doses of rituximab IV over approximately 3-4 hours once weekly for 4 weeks.

Patients are followed at day 100, at 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-Hodgkin's lymphoma

  o Any B cell
* CD20-positive disease
* Failed prior primary induction therapy
* Meets 1 of the following criteria:

  * Chemotherapy-refractory disease
  * Received at least 3 prior chemotherapy regimens
  * Mantle cell lymphoma
* Eligible for transplantation
* 19 years old and over
* WHO 0-2
* Life expectancy at least 6 months
* Absolute neutrophil count ≥ 1,000/mm^3*
* Platelet count > 50,000/mm^3*
* Hemoglobin > 9.0 g/dL*

  o NOTE: *Unless due to lymphomatous involvement of the bone marrow
* Fertile patients must use 2 methods of effective contraception

Exclusion Criteria:

* No history of T-cell lymphoma
* Not pregnant or nursing
* No other concurrent serious disease or condition that would preclude study participation

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2002-05-08 (Actual); Primary Completion 2005-11-01 (Actual); Study Completion 2015-03-12 (Actual)

PRIMARY OUTCOMES:
evaluation of the relationship between levels of sCD20 in the blood of patients with non-Hodgkin's lymphoma pre and post rituximab/BEAM/autologous peripheral blood progenitor cell transplantation (PBPCT) as they relate to clinical outcomes. | pre and post transplant
  To evaluate levels of soluble CD20 antigen (sCD20) in the blood of patients with non-Hodgkin's lymphoma pre and post rituximab/BEAM/autologous hematopoietic stem cell transplantation (AHSCT), and to examine the effect of changes in levels of sCD20 with clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Bociek, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Eppley Cancer Center, Omaha, Nebraska, United States